CLINICAL TRIAL: NCT06281041
Title: Antiplatelet Agents in Patients With Intermediate Coronary Artery Stenosis and Negative Fractional Flow Reserve
Brief Title: Nationwide Cohort Study of Antiplatelet Agents as Primary Prevention
Acronym: NHIS
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Associate Professor, Samsung Medical Center
Other Study IDs: NHIS20240220
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Coronary artery stenosis; Antiplatelet agent; Fractional flow reserve; Prognosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Platelet Aggregation Inhibitors; Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antiplatelet agents: Among patients with intermediate coronary artery stenosis (50-70% diameter stenosis by quantitative coronary angiography) but who did not undergo PCI based on negative FFR, those who were taking antiplatelet agents (aspirin or clopidogrel) are classified into this group.
  Interventions: Drug: Antiplatelet Agents
- No antiplatelet agents: Among patients with intermediate coronary artery stenosis (50-70% diameter stenosis by quantitative coronary angiography) but who did not undergo PCI based on negative FFR, those who were not taking antiplatelet agents (aspirin or clopidogrel) are classified into this group.

INTERVENTIONS:
Drug: Antiplatelet Agents — Aspirin or clopidogrel
  Other Names: aspirin; clopidogrel
  Groups: Antiplatelet agents

SUMMARY:
There is no specific recommendation regarding pharmacologic treatment as primary prevention for patients with intermediate coronary artery stenosis whose revascularization was deferred based on negative fractional flow reserve (FFR).

Current nationwide cohort study conducted using Korean National Health Insurance Service database evaluated the safety and efficacy of antiplatelet therapy in patients with intermediate coronary artery stenosis with deferred revascularization based on negative FFR (FFR>0.80).

DETAILED DESCRIPTION:
This study was nationwide cohort study conducted using Korean National Health Insurance Service database. From 2013 to 2020, reimbursement criteria of FFR were patients with no previous evidence of myocardial ischemia and intermediate coronary artery stenosis (50-70%). Patients who were evaluated by coronary angiography and FFR but did not undergo revascularization were selected and classified according to the use of antiplatelet agents after index procedure. Patients with previous history of atherosclerotic cardiovascular disease were excluded. Eligible patients were matched using propensity score in a 1:1 ratio. Primary efficacy outcome was major adverse cardiac and cerebrovascular events a composite of all-cause death, myocardial infarction, unplanned revascularization, and stroke at 5-year. Primary safety outcome was gastrointestinal bleeding, regardless of the need of transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 50-70% intermediate stenosis by quantitative coronary angiography in a vessel greater than 2.5 mm
* Patients who underwent invasive coronary angiography and FFR measurement
* Patients whose revascularization was deferred based on FFR>0.80

Exclusion Criteria:

* Patients who underween FFR measurement after expansion of reimbursement criteria of FFR (since 2021)
* Patients with history of any bleeding with blood transfusion
* Patients with use of non-vitamin K antagonist oral anticoagulants (NOAC) or warfarin
* Patients with previous atherosclerotic cardiovascular disease
* Patients with already on antiplatelet agents including dual antiplatelet agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2013 to 2020, the use of FFR has been reimbursed by insurance criteria for patients with 50-70% intermediate stenosis by quantitative coronary angiography in a vessel greater than 2.5 mm in the absence of prior evidence of inducible myocardial ischemia by non-invasive tests. The current study included participants who underwent FFR but did not receive revascularization, meaning that they had 50-70% intermediate stenosis and revascularization was deferred based on negative FFR between 2013 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4657 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | at 5 years from index procedure
  Primaey efficacy ouotcome (MACCE, a composite of all-cause death, myocardial infarction, unplanned revascularization, and stroke)
Gastrointestinal bleeding | at 5 years from index procedure
  Primary safety outcome (any gastrointestinal bleeding, regardless of the need of transfusion)

SECONDARY OUTCOMES:
All-cause death | at 5 years from index procedure
  All-cause death which was obtained from death certification collected by Statistics Korea at the Ministry of Strategy and Finance of South Korea.
Myocardial infarction | at 5 years from index procedure
  Myocardial infarction is defined as presence of the diagnostic codes (ICD-10 I21, I22) in the primary position during hospitalization
Unplanned revascularization | at 5 years from index procedure
  Percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) after index hospitalization
Stroke | at 5 years from index procedure
  Stroke is defined as ischemic stroke (ICD-10 I63, I64) or intracranial hemorrhage (ICD-10 I60-62), combined with the codes of diagnostic brain imaging.
Major bleeding | at 5 years from index procedure
  Major bleeding is defined as a composite of intracranial bleeding or gastrointestinal bleeding with documented transfusion.
Gastrointestinal bleeding necessitated hospitalization without documented transfusion | at 5 years from index procedure
  Gastrointestinal bleeding necessitated hospitalization without documented transfusion
Intracranial hemorrhage | at 5 years from index procedure
  Intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center; Danbee Kang, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Chonnam National University Medical School, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No
This is National Helath Insurance Data Analysis. therefore, sharing the original patient-level data is not possible under regulation by Korean Govenment.